CLINICAL TRIAL: NCT02876926
Title: Exploring Use of a Real-time, Remote Monitoring and Follow-up System for Home-based, HIV Self-testing Among High-risk Men Who Have Sex With Men (MSM)
Brief Title: Evaluating a Real-Time, Remote Monitoring System for Home-Based HIV Testing
Acronym: (eTEST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Tyler Wray, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1508001315
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: HIV
Keywords: HIV testing; Self-testing; Counseling; Referral
MeSH Terms: interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- "Enhanced" home-based testing (Experimental): These participants will download a study-specific smartphone app ("eTEST"), and receive home-based HIV test kits in the mail every 3 months. These kits will have been fit with sensors that enable remote detection of when the kit was opened. Qualified HIV test counselors (QHTC) will then follow up with these participants within 24 hours of receiving notification that the test has been opened to conduct routine counseling, offer referrals for other services, and connect those with reactive results with follow-up care.
  Interventions: Behavioral: "Smart" home-based test for HIV
- Home-based testing alone (Active Comparator): These participants will receive a typical home-based test for HIV in the mail every 3 months, but no phone-based follow-up will be provided.
  Interventions: Behavioral: Home-based testing only
- Reminders for clinic-based testing (Sham Comparator): Participants in this condition will receive a letter in the mail every 3 months reminding them to be tested at a local clinic for free.
  Interventions: Behavioral: Reminder letters for clinic-based testing

INTERVENTIONS:
Behavioral: "Smart" home-based test for HIV — A standard home-based HIV test kit, fit with a Bluetooth low energy beacon to allow remote monitoring.
  Arms: "Enhanced" home-based testing
Behavioral: Home-based testing only — A standard home-based HIV test kit.
  Arms: Home-based testing alone
Behavioral: Reminder letters for clinic-based testing — Letters reminding patients to get tested at a free clinic location
  Arms: Reminders for clinic-based testing

SUMMARY:
This study explores whether offering follow-up counseling and referral over the phone after using a home-based HIV test increases rates of ever and repeat testing, compared with home-based testing with no follow-up (HBST alone) or mailing reminders for clinic-based testing.

ELIGIBILITY:
Inclusion Criteria:

* Sex with a partner met online in the past year
* Anal sex (either insertive or receptive) with a casual male partner in the past 6 months without using condoms or pre-exposure prophylaxis
* Own a smartphone (iOS or Android) with a service contract and data plan
* Have a stable address where mail can be received
* Speak English fluently

Exclusion Criteria:

* Having tested for HIV in the last year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Enhanced" Home-based Testing | Home-based Testing Alone | Reminders for Clinic-based Testing
Started | 21 | 22 | 22
Completed | 3 | 3 | 2
Not Completed | 18 | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Enhanced" Home-based Testing | Home-based Testing Alone | Reminders for Clinic-based Testing | Total
Number analyzed (Participants) | 21 | 22 | 22 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 22 | 22 | 65
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (13.9) | 35.8 (16.3) | 35.5 (15.2) | 35.2 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 21 | 22 | 22 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 7
  White | 16 | 20 | 14 | 50
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 22 | 22 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received HIV Testing
Description: Count of the number of participants who reported receiving HIV testing.
Time Frame: Up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | "Enhanced" Home-based Testing | Home-based Testing Alone | Reminders for Clinic-based Testing
Number analyzed (Participants) | 21 | 22 | 22
Participants | 21 | 22 | 16

2. Primary Outcome: Number of Participants Who Reported Having Been Referred for Pre-exposure Prophylaxis
Description: Count of the number of participants who reported receiving a referral for pre-exposure prophylaxis from a counselor or medical professional.
Time Frame: Up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | "Enhanced" Home-based Testing | Home-based Testing Alone | Reminders for Clinic-based Testing
Number analyzed (Participants) | 21 | 22 | 22
Participants | 8 | 2 | 3

3. Primary Outcome: Number of Participants Who Reported Having Actually Received a Prescription for Pre-exposure Prophylaxis
Description: Count of the number of participants who reported actually having received a prescription for pre-exposure prophylaxis after having been referred by a medical professional.
Time Frame: Up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | "Enhanced" Home-based Testing | Home-based Testing Alone | Reminders for Clinic-based Testing
Number analyzed (Participants) | 21 | 22 | 22
Participants | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected monthly over the course of the 7-month study period.
Arm/Group | "Enhanced" Home-based Testing | Home-based Testing Alone | Reminders for Clinic-based Testing
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02876926/SAP_000.pdf
  • Study Protocol (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02876926/Prot_001.pdf